CLINICAL TRIAL: NCT02475824
Title: A Randomized Comparison of Midazolam With Meperidine and Dexmedetomidine Versus Midazolam With Meperidine and Propofol for Sedation During ERCP
Brief Title: Midazolam With Meperidine and Dexmedetomidine vs. Midazolam With Meperidine and Propofol for Sedation During ERCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dankook University (Other)
Responsible Party: Principal Investigator, Jun Ho Choi, Assistant professor, Dankook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DankookU
Record Dates: First submitted 2015-06-14; First posted 2015-06-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Complication
Keywords: ERCP; Sedation; safety
MeSH Terms: interventions — Midazolam; Meperidine; Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MMD arm (Experimental): Both midazolam® (0.05 mg/kg, 30% reduction for patients if age ≥70 or ASA class III-IV; Bukwang Pharm Co., Seoul, Republic of Korea) and meperidine (50mg. 25mg for patients aged ≥70 years; pethidine HCL, Hana Pharm Co., Seoul, Republic of Korea) are given intravenously at the initiation of sedation. In addition, a continuous IV infusion of dexmedetomidine (1ug/kg/h, Precedex; Hospira, Seoul, Republic of Korea) is administered 15 min before the ERCP till complete procedure
  Interventions: Drug: Midazolam®; Drug: "Meperidine" (pethidine®); Drug: Dexmedetomidine (Precedex®)
- BPS arm (Active Comparator): IV bolus dose of midazolam® (0.06mg/kg, 50% reduction for patients if age ≥70 or ASA class III-IV; Bukwang Pharm Co., Seoul, Republic of Korea) and meperidine (50mg. 25mg for patients aged ≥70 years; pethidine HCL, Hana Pharm Co., Seoul, Republic of Korea). Repeated doses of 10-20 mg propofol® are titrated to achieve the target level of sedation. 0.9% NaCl 1μg/Kg•hr IV continuous infusion, initiated 15 min before the procedure (ERCP) till complete procedure
  Interventions: Drug: Midazolam®; Drug: "Meperidine" (pethidine®); Drug: Propofol®

INTERVENTIONS:
Drug: Midazolam® — midazolam (0.05 mg/kg, 30% reduction for patients if age ≥70 or ASA class III-IV; Bukwang Pharm Co., Seoul, Republic of Korea)
  Other Names: Midazolam
Drug: "Meperidine" (pethidine®) — Meperidine (50mg. 25mg for patients aged ≥70 years; pethidine HCL, Hana Pharm Co., Seoul, Republic of Korea).
  Other Names: meperidine
Drug: Propofol® — Repeated doses of 10-20 mg propofol are titrated to achieve the target level of sedation.
  Other Names: Propofol
  Arms: BPS arm
Drug: Dexmedetomidine (Precedex®) — Dexmedetomidine (1μg/kg/h, Precedex; Hospira, Seoul, Republic of Korea) or the same volume of normal saline were administered in the MMD and midazolam-meperidine group
  Other Names: Dexmedetomidine
  Arms: MMD arm

SUMMARY:
This is a single-center, prospective, randomized, double-blinded study of consecutive patients referred for ERCP. A recent study suggested that the addition of dexmedetomidine to the midazolam-meperidine regimen (MMD)provided better sedative efficacy and a superior safety profile during ERCP compared with a midazolam-meperidine regimen. Further study is warranted to compare an MMD regimen with propofol-based regimen.

Randomization is performed by use of a computer-generated random allocations in a ratio of 1:1 in balanced blocks of 4. A separate sedating nurse, who don't participate in the study, is the only person with knowledge of the sedation regimen. This separate nurse repeated the injection of propofol and completed questionnaires.

DETAILED DESCRIPTION:
Study design This is a single-center, prospective, randomized, double-blinded study of consecutive patients referred for ERCP. Randomization is performed by use of a computer-generated random allocations in a ratio of 1:1 in balanced blocks of 4. A separate sedating nurse, who don't participate in the study, is the only person with knowledge of the sedation regimen. This separate nurse repeated the injection of propofol and completed questionnaires.

Inclusion criteria include consecutive patients who are scheduled for ERCP and those are aged 18-80 years. (ASA class I-III) Exclusion criteria are as follows;

1) patient age < 18years, 2) pregnancy, 3) American Society of Anesthesiology (ASA) physical status class IV, V, 4) history of allergies to drug used, 6) history of complications with previous sedation, 5) hypoxemia (baseline SaO2) <90%, 6) hypotension (baseline systolic blood pressure <90mmHg), 7) severe bradycardia (heart rate <50/min) and/or brady-dysrhythmias (e.g. advanced heart block), 8) impaired ventricular function (left ventricular ejection fraction <30%), 9) baseline respiratory rate >25 or <10 breaths/min, and 10) inability to provide informed consent. Patients are excluded from the final analysis if the procedure is terminated early or abandoned for anatomical reasons (i.e., duodenal obstruction or gastrectomy).

Sedation protocols After randomization patients are allocated to group 1 or 2, and prepared for endoscopy.

All sedatives and analgesics used for the study are administered by trained sedative nurse under endoscopist supervision. All participants receive an IV bolus dose of midazolam (0.06mg/kg, 50% reduction for patients if age ≥70 or ASA class III-IV; Bukwang Pharm Co., Seoul, Republic of Korea) and meperidine (50mg. 25mg for patients aged ≥70 years; pethidine HCL, Hana Pharm Co., Seoul, Republic of Korea). Repeated doses of 10-20 mg propofol are titrated to achieve the target level of sedation. Maintenance of sedation is achieved with repeated doses of 5 to 20 mg propofol. The total dosage of propofol (including additional doses) is limited by lower and upper bounds of 10mg and 100mg, respectively. The target level of sedation is moderate sedation based on the ASA levels.

For the patients allocated to the midazolam-meperidine-dexmedetomidine (MMD) group, both midazolam (0.05 mg/kg, 30% reduction for patients if age ≥70 or ASA class III-IV; Bukwang Pharm Co., Seoul, Republic of Korea) and meperidine (50mg. 25mg for patients aged ≥70 years; pethidine HCL, Hana Pharm Co., Seoul, Republic of Korea) are given intravenously at the initiation of sedation. In addition, a continuous IV infusion of dexmedetomidine (1ug/kg/h, Precedex; Hospira, Seoul, Republic of Korea) is administered 15 min before the ERCP till complete the procedure. Thereafter, repeated doses of 1 to 2 mg midazolam are administered to maintain a moderate level of sedation. For the patients allocated to the midazolam-meperidine-propofol (BPS) group, both midazolam and meperidine are given at the initiation of sedation in the same manner as in the MMD group.

Thereafter, repeated doses of 10-20 mg propofol are titrated to achieve the target level of sedation. Maintenance of sedation is achieved with repeated doses of 5 to 20 mg propofol. The total dosage of propofol (including additional doses) is limited by lower and upper bounds of 10mg and 100mg, respectively. The target level of sedation is moderate sedation based on the ASA levels.

Medications and monitoring Intranasal supplemental oxygen (2L/min) is provided to all participants at the initiation of sedation. Heart rate, electrocardiogram, peripheral oxygen saturation (SaO2), respiratory rate, and end-tidal carbon dioxide (EtCo2) are constantly monitored. Non-invasive blood pressure (NIBP) is automatically measured at 3-minute intervals. Sedation level is assessed and recorded every 3 minutes throughout the procedure with the Modified Observer's Assessment of Alertness and Sedation (MOAA/S). Patients are considered to be oversedated at MOAA/S score 1.

MOAA/S, Modified Observe's Assessment of Alertness and Sedation: 5-responds readily to name spoken in normal tone, 4-lethargic response to name spoken in normal tone, 3-responds only after name is called loudly and/or repeatedly, 2-responds only after mild prodding or shaking, 1-does not respond to mild prodding or shaking, 0-does not respond to noxious stimulus.

If hypoxemia (SpO2<90%) is observed during sedation in either group, O2 supplementation is increased by 2L/min until oxygen saturation is restored. If the SpO2 dropped to < 85% for >30 sec, despite patient stimulation and interruption of sedatives and jaw thrust maneuver, an antagonist to midazolam (flumazenil) could be injected and the procedure is interrupted until normalization of oxygen saturation occurred again.

During recovery, the patient's vital signs (NIBP, SpO2, heart rate), sedation level (Gillham scale), and speed of recovery (modified Aldrete score) are recorded at 5-minute intervals until discharge from the recovery room.

Gillham sedation scale; 1-awake and anxious, 2-awake not anxious, 3-speech slurred, 4-eyes closed, responds to speech, 5-eye closed, responds to shaking, 6-unresponsive.

Outcome measurements and definitions The primary endpoint of the study is the rates of cardiopulmonary complications and the frequency of interruption of the ERCP procedures because of complications included (1) hypoxemia (pulse oximeter oxygen saturation below 90% on supplemental oxygen), (2) hypotension (systolic blood pressure below 90 mmHg), (3) bradycardia (heart rate below 50 beats/min). Procedure quality is evaluated based on therapeutic procedure outcomes, including technical success and total procedure time, and procedure-related adverse events. If transient interruptions of the procedure occurred because of sedation-related complications, that time is subtracted from the procedure time.

The endoscopist, blinded to the method of sedation, The secondary endpoints are the ease of ERCP performance, speed of recovery, and patient satisfaction with sedation.

At the end of the procedure, the ease of performance of ERCP is evaluated by the endoscopist using structured questionnaires.

If full recovery is confirmed in the inpatient setting, patient satisfaction with sedation and pain intensity during ERCP are assessed by another independent assistant using a 10-cm VAS scale (0=no pain/no satisfaction, 10=worst pain/full satisfaction)

ELIGIBILITY:
Inclusion Criteria:

* Those who are scheduled for ERCPs
* aged 18 to 80 years
* American Society of Anesthesiologists (ASA) classification I to III

Exclusion Criteria:

* ASA IV and V
* History of allergies to drug used
* refuse to participate the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
the rates of cardiopulmonary complications | From start point of the procedure(ERCP) to 60 minutes after the procedure
  respiratory depression (≤10 breaths/min); desaturation (SaO2<90% with no recovery against a verbal stimulus or jaw extension); hypotension (systolic blood pressure <90mmHg or 20% reduction from baseline mean blood pressure

SECONDARY OUTCOMES:
Sedation efficacy | From start point of the procedure(ERCP) to 1 hour after the procedure
  Modified Observe's Assessment of Alertness and Sedation: 5-responds readily to name spoken in normal tone, 4-lethargic response to name spoken in normal tone, 3-responds only after name is called loudly and/or repeatedly, 2-responds only after mild prodding or shaking, 1-does not respond to mild prodding or shaking, 0-does not respond to noxious stimulus.
procedural satisfaction | From start point of the procedure(ERCP) to 1 day after the procedure
  respective visual analog scale (VAS; 0=no pain/ no satisfaction, 10=worst pain imaginable/full satisfaction
Speed of recovery | From start point of the procedure(ERCP) to 1 hour after the procedure
  speed of recovery (modified Aldrete score) are recorded at 5-minute intervals until discharge from the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ho Choi, MD, Principal Investigator — Dankook University
Locations (1):
- Dankook University College of Medicine, Cheonan, Chungcheongnam-do, South Korea